CLINICAL TRIAL: NCT05559060
Title: Comorbidities of Epilepsy(Cognitive and Psychiatric Dysfunction)
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Hasnaa Abdallah, Resident doctor, Assiut University
Other Study IDs: Comrbidities of epilepsy
Record Dates: First submitted 2022-09-24; First posted 2022-09-29 (Actual); Last update posted 2022-09-29 (Actual); Status verified 2022-09

CONDITIONS: Epilepsy
MeSH Terms: conditions — Epilepsy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Epilepsy is the second commonest chronic neurological disorder in developed countries ,comorbidity refers to the co-occurrence of two conditions with greater frequency than found in the general population

ELIGIBILITY:
Inclusion Criteria:

Patients with primary epilepsy. Aged above 18 years old.

Exclusion Criteria:

* patient diagnosed as secondary epilepsy or epilepsy syndromes

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects included will be chosen from epilepsy clinic and neurology department at assiut University hospital
Sampling Method: Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2022-09 (Estimated); Primary Completion 2023-05 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Find out comorbidities of epilesy and its treatment | 1 year

IPD SHARING:
Plan to Share IPD: Undecided